CLINICAL TRIAL: NCT05710185
Title: Deucravacitinib for the Treatment of Palmoplantar Pustulosis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor terminated funding
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Arash Mostaghimi, M.D., M.P.A., M.P.H., Associate Professor of Dermatology, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023P000194
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Palmoplantar Pustulosis
MeSH Terms: conditions — Psoriasis | interventions — deucravacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Subjects with Palmoplantar pustulosis (Experimental): All participants will receive deucravacitinib 6 mg daily for 24 weeks, with study visits every 4 weeks.
  Interventions: Drug: Deucravacitinib

INTERVENTIONS:
Drug: Deucravacitinib — See arm/group description

SUMMARY:
A prospective, single-arm, open-label trial of deucravacitinib 6 mg daily in patients with PPP. All participants will receive deucravacitinib 6 mg daily for 24 weeks, with study visits every 4 weeks.

DETAILED DESCRIPTION:
Objectives:

1. Evaluate the efficacy of deucravacitinib in adults with PPP
2. Evaluate the impact of deucravacitinib on quality of life in adults with PPP
3. Evaluate the safety of deucravacitinib Primary Endpoint: • Proportion of participants who achieve a ppPASI-50 response, or at least 50% improvement in ppPASI score, at 16 weeks Secondary Endpoints: • Proportion of participants who achieve at least 50% improvement in the palmoplantar pustular psoriasis area and severity index (ppPASI-50) at 24 weeks

   * Frequency of participants with adverse events
   * Change from baseline in the Dermatology Quality of Life Index
   * Change from baseline in ppPASI
   * Percentage of patients who achieved a static Physician's Global Assessment score of 0/1
   * Change from baseline in the EQ-5D VAS score
   * Change from baseline in itch VAS
   * Change from baseline in pain VAS Inclusion Criteria: • Adults aged 18 years of age and older
   * Dermatologist confirmed diagnosis of PPP for at least 6 months
   * Moderate-severe PPP, defined as a ppPASI > 12
   * Inadequate response to topical therapy and a candidate for systemic or phototherapy
   * Willing to discontinue current topical and/or systemic PPP treatments, except for OTC emollients Exclusion Criteria: • Participants with other immune-mediated conditions requiring concurrent systemic immunosuppressant treatments
   * Current/recent administration of PPP-specific medications including:

     * Rituximab within 6 months of the baseline visit
     * Biologics within 12 weeks of baseline visit
     * Systemic steroids, oral immunosuppressants (azathioprine, cyclosporine, methotrexate, mycophenolate mofetil, tacrolimus), oral retinoids (acitretin, isotretinoin), apremilast, or dapsone within 4 weeks of baseline visit
     * Phototherapy within 4 weeks of baseline visit
     * Prescription topical medications (including calcineurin inhibitors, crisaborole, retinoids, steroids, tar, vitamin D analogs) within 2 weeks of baseline visit
   * History of active infection and/or febrile illness within 7 days; or infection requiring antibiotic treatment within 30 days; or serious infection requiring hospitalization and/or IV antibiotics within 90 days
   * Evidence of other infection including:

     * Active or untreated latent tuberculosis, defined as radiographic or laboratory evidence of active TB or positive quantiferon or PPD, unless the subject has completed the recommended treatment
     * Human immunodeficiency virus infection (positive HIV antibody)
     * Active hepatitis B
     * Active hepatitis C
   * Evidence of clinically significant laboratory abnormality including:

     * Absolute WBC count < 3000/mm3
     * Platelet count < 100,000/mm3
     * Hemoglobin < 9.0 g/dl
     * ALT or AST > 3 times the upper limit of normal
   * History of cancer within the past 5 years, excluding treated non-melanoma skin cancer (basal cell carcinoma, squamous cell carcinoma)
   * Other uncontrolled chronic medical condition that may interfere with a patient's ability to participate in the clinical trial
   * Major surgery within 4 weeks of baseline visit
   * Receipt of live vaccine within 8 weeks of baseline visit
   * Pregnant or breastfeeding individuals
   * Inability to comply with any of the study procedures
   * Individuals who are incarcerated or compulsory detained Sample Size: A modified Simon's two-stage design will be used to maximize the safety and efficiency of this clinical trial in an orphan disease. In the first stage, 8 patients will be accrued. If 2 or fewer patients achieve a ppPASI-50 in these 8 patients, the study will be stopped. Otherwise, 10 additional patients will be accrued for a total of 18.

Analysis Plan: Descriptive statistics will be used to characterize the study population, including demographics, disease characteristics and previous treatments. For the primary outcome, the percentage of participants who achieve a ppPASI-50 response, or at least 50% improvement in ppPASI score, at 16 weeks, the response rate with a 95% CI will be calculated. For all secondary endpoints, summary and descriptive statistics will be used as appropriate , including number of observations, calculation of mean/median, standard deviation range and 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* • Adults aged 18 years of age and older

  * Dermatologist confirmed diagnosis of PPP for at least 6 months
  * Moderate-severe PPP, defined as a ppPASI > 12
  * Inadequate response to topical therapy and a candidate for systemic or phototherapy
  * Willing to discontinue current topical and/or systemic PPP treatments, except for OTC emollients

Exclusion Criteria:

* • Participants with other immune-mediated conditions requiring concurrent systemic immunosuppressant treatments

  * Current/recent administration of PPP-specific medications including:

    * Rituximab within 6 months of the baseline visit
    * Biologics within 12 weeks of baseline visit
    * Systemic steroids, oral immunosuppressants (azathioprine, cyclosporine, methotrexate, mycophenolate mofetil, tacrolimus), oral retinoids (acitretin, isotretinoin), apremilast, or dapsone within 4 weeks of baseline visit
    * Phototherapy within 4 weeks of baseline visit
    * Prescription topical medications (including calcineurin inhibitors, crisaborole, retinoids, steroids, tar, vitamin D analogs) within 2 weeks of baseline visit
  * History of active infection and/or febrile illness within 7 days; or infection requiring antibiotic treatment within 30 days; or serious infection requiring hospitalization and/or IV antibiotics within 90 days
  * Evidence of other infection including:

    * Active or untreated latent tuberculosis, defined as radiographic or laboratory evidence of active TB or positive quantiferon or PPD, unless the subject has completed the recommended treatment
    * Human immunodeficiency virus infection (positive HIV antibody)
    * Active hepatitis B
    * Active hepatitis C
  * Evidence of clinically significant laboratory abnormality including:

    * Absolute WBC count < 3000/mm3
    * Platelet count < 100,000/mm3
    * Hemoglobin < 9.0 g/dl
    * ALT or AST > 3 times the upper limit of normal
  * History of cancer within the past 5 years, excluding treated non-melanoma skin cancer (basal cell carcinoma, squamous cell carcinoma)
  * Other uncontrolled chronic medical condition that may interfere with a patient's ability to participate in the clinical trial
  * Major surgery within 4 weeks of baseline visit
  * Receipt of live vaccine within 8 weeks of baseline visit
  * Pregnant or breastfeeding individuals
  * Inability to comply with any of the study procedures
  * Individuals who are incarcerated or compulsory detained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Pennsylvania, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subjects with Palmoplantar pustulosis
Started | 3
Completed | 1
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Subjects With Palmoplantar Pustulosis
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Achieve a ppPASI-50 Response, or at Least 50% Improvement in ppPASI Score
Description: The ppPASI is the most commonly used disease severity measure use in palmoplantar pustulosis clinic trials. The ppPASI is composed of subscores of erythema (E), pustules/vesicles (P), desquamation/scales (D) on the left (L) and right (R) palm (P) and sole (S) respectively. The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects with Palmoplantar pustulosis
Number analyzed (Participants) | 2
Participants | 0
Statistical Analysis 1: Comparison: Subjects with Palmoplantar pustulosis; Test type: Other; It was a descriptive study

2. Primary Outcome: Proportion of Participants Who Achieve a ppPASI-50 Response, or at Least 50% Improvement in ppPASI Score
Description: The ppPASI is the most commonly used disease severity measure use in palmoplantar pustulosis clinic trials. The ppPASI is composed of subscores of erythema (E), pustules/vesicles (P), desquamation/scales (D) on the left (L) and right (R) palm (P) and sole (S) respectively. The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity.
  This second Primary Outcome was added by administrative error since the study only has one Primary Outcome Measure. Hence, the outcome and results are a duplication of the outcome measure reported, and this one was left incomplete in the previous results reporting submission.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects with Palmoplantar pustulosis
Number analyzed (Participants) | 2
Participants | 0

3. Secondary Outcome: Change From Baseline in the Dermatology Quality Life Index (DLQI)
Description: The DLQI is a dermatology-specific quality of life instrument to measure the impact of skin disease on different aspects of health-related quality of life. The questionnaire contains 10 questions, each scored on a 4-point Likert scale. The DLQI is calculated by adding the score of each question, resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. A score higher than 10 indicates that the patient's life is being severely affected by their skin disease.
Time Frame: Week 16, Week 24
Reporting Status: Not Posted

4. Secondary Outcome: Change From Baseline in ppPASI
Description: as for outcome 1
Time Frame: Week 16, Week 24
Reporting Status: Not Posted

5. Secondary Outcome: Percentage of Patient Who Achieve a Physicians Global Assessment Score of 0 or 1
Description: The physician's global assessment is a widely used outcome measure that relies on physician visual assessment of disease severity. The static PGA determines psoriasis severity at a single point in time, without taking the baseline disease condition into clear (0), almost clear (1), mild (2), moderate (3), severe (4).
Time Frame: Week 16, Week 24
Reporting Status: Not Posted

6. Secondary Outcome: Change From Baseline in EQ-5D VAS
Description: The EQ-5D is a validated, reliable, and responsive instrument widely used in clinical trials where respondents rate their health in each of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety depression. EQ-5D questionnaire also includes a Visual Analog Scale (VAS), by which respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).
Time Frame: Week 16, Week 24
Reporting Status: Not Posted

7. Secondary Outcome: Change From Baseline in the Itch Visual Analogue Scale (Itch-VAS)
Description: The VAS-itch is a 10 cm line on which patients mark their pruritus intensity on a scale from "no itch" (0 points) to "worst imaginable itch" (10 points). The VAS-itch can be interpreted as 0 - < 3 points represents mild pruritus, ≥ 3 - 7 points moderate pruritus, ≥ 7 - 9 points severe pruritus, and ≥ 9 points severe pruritus
Time Frame: Week 16, Week 24
Reporting Status: Not Posted

8. Secondary Outcome: Change From Baseline in the Pain Visual Analogue Scale (Pain-VAS)
Description: The VAS-pain is a 10 cm line on which patients mark their pain on a scale from "no no" (0 points) to "worst imaginable pain" (100 points). The following cut points on the pain VAS have been recommended pain: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75 - 100 mm)
Time Frame: Week 16, 24
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Subjects with Palmoplantar pustulosis
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects with Palmoplantar pustulosis (N=3)
Infection (Infections and infestations) | 1 (1) — Ear infection requiring antibiotic treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/85/NCT05710185/Prot_SAP_001.pdf